CLINICAL TRIAL: NCT01849133
Title: Randomized Clinical Trial: Comparison Between Quadrantectomy Followed by External Fractionated Radiotherapy and Quadrantectomy Associated With Intraoperative Radiotherapy in Women >= 48 Years of Age Affected by Early-stage Breast Carcinoma.
Brief Title: Randomized Trial on Intraoperative Radiotherapy Full Dose Vs External Radiotherapy
Acronym: ELIOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEO S65/500
Record Dates: First submitted 2013-05-05; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Carcinoma Breast
Keywords: Breast cancer; conservative surgery; intraoperative radiation therapy; mobile linear accelerator
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ELIOT (Experimental): intraoperative radiotherapy
  Interventions: Radiation: intraoperative radiotherapy
- EXTERNAL RT (Active Comparator): external fractionated radiotherapy
  Interventions: Radiation: external fractionated radiotherapy

INTERVENTIONS:
Radiation: external fractionated radiotherapy — conventional external beam radiotherapy
  Arms: EXTERNAL RT
Radiation: intraoperative radiotherapy — Intraoperative radiotherapy (IORT). Total delivered dose 21Gy (Gray), 90% isodose
  Arms: ELIOT

SUMMARY:
The purpose of this study is to investigate the efficacy of exclusive intraoperative radiation therapy after conserving surgery in early-stage breast cancer compared with whole breast radiotherapy. The primary outcome was the rate of ipsilateral true recurrence ( any recurrence at or close to primary tumor bed) and new ipsilateral tumors ( any recurrence occurring in quadrants other than the previous one) and the recurrence free survival.

DETAILED DESCRIPTION:
The ELIOT trial is a prospective single center randomised phase III trial which compared intraoperative radiotherapy with electrons to the tumor bed with conventional scheme of whole breast external beam radiotherapy. Patients were randomly allocated to intraoperative radiotherapy group or external radiotherapy group in a 1:1 ratio.

The rationale for providing partial breast irradiation to the tumor bed lies on the patterns of ipsilateral breast tumor relapse reported in Literature. In fact, the majority of recurrences occur close to the tumor bed. Several randomized trials of breast conserving surgery with or without whole breast radiotherapy showed that in 75-90% of cases recurrences were at the site of original primary tumor. In this context, limiting irradiation to the tumor bed may result in a similar local control as whole breast irradiation, provided that patients are properly selected.

The intraoperative treatment was delivered with a mobile miniaturized accelerator, located in the operating room, while for external radiotherapy a 6 MV linear accelerator was used. The surgical technique to perform ELIOT has been standardized in every step. The breast gland is prepared by separating it from the subcutaneous tissue and the underlying pectoralis muscle and by restoring the continuity of the surgical breach after having protected the thoracic wall by lead and aluminium disks to optimize the delivered dose. The linear accelerator delivers electrons at variable energy, ranging from 3 to 9 MeV: the proper electron energy is chosen according to the target thickness. Collimation is achieved by hard-docking system, consisting of 5 mm thick high- quality polymethyl methacrylate round applicators of 4 to 10 -cm diameter.

For radiation protection a primary beam stopper and mobile 1.5 cm thick lead shields are provided. The prescribed dose was 21 Gy at the 90% isodose. After delivery of the radiation dose, the applicator and the disk were removed and the gland is reconstructed again.

In the conventional arm of the study, the external beam radiotherapy is given after the full recovery from the surgical excision. All patients undergo virtual simulation including a treatment-planning CT scan. The clinical target volume is defined to extend to 5 mm below the skin surface and include breast parenchyma down to the deep fascia, but not including the underlying muscle and rib cage. The irradiated volume should extend medially to the midline, laterally to the mid axillary line and inferiorly to 1-2 cm below the level of intra-mammary fold and superiorly to the suprasternal notch. Using BEV, the blocks are used to shield as much heart and lung as possible without compromising the PTV.

Treatment is delivered by a pair of tangential fields with wedges as necessary. The prescribed dose to the whole-breast was 50 Gy delivered in 2 Gy fraction over 5 weeks with a 6 -megavolt linear accelerator followed by a sequential boost of 10 Gy to the tumor bed with electrons. A PTV dose homogeneity of -5% + 7% as recommended by ICRU (International Commission on Radiation Units and Measurements) report no 50.

Patients were followed up with at least 6-month clinical examination up to 5 years and then every 8 months thereafter. Annual mammogram was performed .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 48 and < 75
* Clinical mammographic/ultrasound diagnosis of unicentric carcinoma, with ultrasound diameter ≤2.5 cm. Advisable, but not mandatory, the execution of mammoscintigraphy with MDP-99mTc (Methyl diphosphonate technetium-99m) : this procedure allows the bone staging and the mapping of eventual multi-focality/multi-centricity of the breast neoplasm.
* No previous therapy (biopsy included) for breast cancer in other Institutions.
* Patients with non-palpable lesions will undergo preoperative centering and stereotactic and/or ultrasound-guided cytology (the execution of this last procedure is not mandatory).
* Adequate information to the patient and informed consent.

Exclusion Criteria:

* Ductal or lobular non-infiltrating carcinoma.
* Paget disease.
* Tumor in close proximity to the skin.
* Tumor in the axillary tail.
* Documented multi-centricity/multi-focality of the tumor.
* Patients who underwent excisional biopsy in other Institutions.
* Histology different from carcinoma.
* Personal anamnesis positive for malignancy (basocellular carcinoma, in situ carcinoma of the cervix, contralateral breast cancer free of disease after 15 years of follow-up excluded).
* General contraindications to regular follow-up or radiotherapy.

Ages: 48 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1305 (Actual)
Dates: Start 2000-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of local relapses | 5 YEARS
  local relapse of disease and ipsilateral second primary

CONTACTS AND LOCATIONS:
Overall Officials: UMBERTO VERONESI, PROF, Study Chair — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Background] Veronesi U, Orecchia R, Luini A, Gatti G, Intra M, Zurrida S, Ivaldi G, Tosi G, Ciocca M, Tosoni A, De Lucia F. A preliminary report of intraoperative radiotherapy (IORT) in limited-stage breast cancers that are conservatively treated. Eur J Cancer. 2001 Nov;37(17):2178-83. doi: 10.1016/s0959-8049(01)00285-4. PMID 11677104
- [Background] Gatzemeier W, Orecchia R, Gatti G, Intra M, Veronesi U. [Intraoperative radiotherapy (IORT) in treatment of breast carcinoma--a new therapeutic alternative within the scope of breast-saving therapy? Current status and future prospects. Report of experiences from the European Institute of Oncology (EIO), Mailand]. Strahlenther Onkol. 2001 Jul;177(7):330-7. doi: 10.1007/pl00002415. German. PMID 11505618
- [Background] Intra M, Gatti G, Luini A, Galimberti V, Veronesi P, Zurrida S, Frasson A, Ciocca M, Orecchia R, Veronesi U. Surgical technique of intraoperative radiotherapy in conservative treatment of limited-stage breast cancer. Arch Surg. 2002 Jun;137(6):737-40. doi: 10.1001/archsurg.137.6.737. PMID 12049547
- [Background] Veronesi U, Gatti G, Luini A, Intra M, Orecchia R, Borgen P, Zelefsky M, McCormick B, Sacchini V. Intraoperative radiation therapy for breast cancer: technical notes. Breast J. 2003 Mar-Apr;9(2):106-12. doi: 10.1046/j.1524-4741.2003.09208.x. PMID 12603383
- [Background] Ciocca M, Orecchia R, Garibaldi C, Rondi E, Luini A, Gatti G, Intra M, Veronesi P, Lazzari R, Tosi G, Veronesi U. In vivo dosimetry using radiochromic films during intraoperative electron beam radiation therapy in early-stage breast cancer. Radiother Oncol. 2003 Dec;69(3):285-9. doi: 10.1016/j.radonc.2003.09.001. PMID 14644488
- [Background] Orecchia R, Ciocca M, Lazzari R, Garibaldi C, Leonardi MC, Luini A, Intra M, Gatti G, Veronesi P, Petit JI, Veronesi U. Intraoperative radiation therapy with electrons (ELIOT) in early-stage breast cancer. Breast. 2003 Dec;12(6):483-90. doi: 10.1016/s0960-9776(03)00156-5. PMID 14659125
- [Background] Veronesi U, Gatti G, Luini A, Intra M, Ciocca M, Sanchez D, Zurrida S, Navarro S, Orecchia R. Full-dose intraoperative radiotherapy with electrons during breast-conserving surgery. Arch Surg. 2003 Nov;138(11):1253-6. doi: 10.1001/archsurg.138.11.1253. PMID 14609877
- [Background] Intra M, Leonardi MC, Gatti G, Vento AR, Ciocca M, Veronesi P, Bassani G, Dos Santos GR, Rodriguez J, Luini A, Orecchia R, Veronesi U. Intraoperative radiotherapy during breast conserving surgery in patients previously treated with radiotherapy for Hodgkin's disease. Tumori. 2004 Jan-Feb;90(1):13-6. doi: 10.1177/030089160409000104. PMID 15143964
- [Background] Intra M, Orecchia R, Veronesi U. Intraoperative radiotherapy: the debate continues. Lancet Oncol. 2004 Jun;5(6):340. doi: 10.1016/S1470-2045(04)01489-5. No abstract available. PMID 15172353
- [Background] Orecchia R, Ciocca M, Tosi G, Franzetti S, Luini A, Gatti G, Veronesi U. Intraoperative electron beam radiotherapy (ELIOT) to the breast: a need for a quality assurance programme. Breast. 2005 Dec;14(6):541-6. doi: 10.1016/j.breast.2005.08.038. Epub 2005 Oct 19. PMID 16242331
- [Background] Intra M, Leonardi C, Luini A, Veronesi P, Gennari R, Gatti G, Ciocca M, Soteldo J, Bassi F, Venturino M, Orecchia R, Veronesi U. Full-dose intraoperative radiotherapy with electrons in breast surgery: broadening the indications. Arch Surg. 2005 Oct;140(10):936-9. doi: 10.1001/archsurg.140.10.936. PMID 16230541
- [Background] Luini A, Orecchia R, Gatti G, Intra M, Ciocca M, Galimberti V, Veronesi P, Santos GR, Gilardi D, Veronesi U. The pilot trial on intraoperative radiotherapy with electrons (ELIOT): update on the results. Breast Cancer Res Treat. 2005 Sep;93(1):55-9. doi: 10.1007/s10549-005-3782-1. PMID 16184459
- [Background] Orecchia R, Luini A, Veronesi P, Ciocca M, Franzetti S, Gatti G, Veronesi U. Electron intraoperative treatment in patients with early-stage breast cancer: data update. Expert Rev Anticancer Ther. 2006 Apr;6(4):605-11. doi: 10.1586/14737140.6.4.605. PMID 16613547
- [Background] Petit JY, Veronesi U, Orecchia R, Luini A, Rey P, Intra M, Didier F, Martella S, Rietjens M, Garusi C, DeLorenzi F, Gatti G, Leon ME, Casadio C. Nipple-sparing mastectomy in association with intra operative radiotherapy (ELIOT): A new type of mastectomy for breast cancer treatment. Breast Cancer Res Treat. 2006 Mar;96(1):47-51. doi: 10.1007/s10549-005-9033-7. Epub 2005 Oct 27. PMID 16261402
- [Background] Calvo FA, Meirino RM, Orecchia R. Intraoperative radiation therapy first part: rationale and techniques. Crit Rev Oncol Hematol. 2006 Aug;59(2):106-15. doi: 10.1016/j.critrevonc.2005.11.004. Epub 2006 Jul 14. PMID 16844383
- [Background] Calvo FA, Meirino RM, Orecchia R. intraoperative radiation therapy part 2. Clinical results. Crit Rev Oncol Hematol. 2006 Aug;59(2):116-27. doi: 10.1016/j.critrevonc.2006.04.004. Epub 2006 Jul 21. PMID 16859922
- [Background] Bernier J, Viale G, Orecchia R, Ballardini B, Richetti A, Bronz L, Franzetti-Pellanda A, Intra M, Veronesi U. Partial irradiation of the breast: Old challenges, new solutions. Breast. 2006 Aug;15(4):466-75. doi: 10.1016/j.breast.2005.11.012. Epub 2006 Jan 24. PMID 16439129
- [Background] Ciocca M, Piazzi V, Lazzari R, Vavassori A, Luini A, Veronesi P, Galimberti V, Intra M, Guido A, Tosi G, Veronesi U, Orecchia R. Real-time in vivo dosimetry using micro-MOSFET detectors during intraoperative electron beam radiation therapy in early-stage breast cancer. Radiother Oncol. 2006 Feb;78(2):213-6. doi: 10.1016/j.radonc.2005.11.011. Epub 2005 Dec 15. PMID 16359743
- [Background] Luini A, Gatti G, Zurrida S, Talakhadze N, Brenelli F, Gilardi D, Paganelli G, Orecchia R, Cassano E, Viale G, Sangalli C, Ballardini B, dos Santos GR, Veronesi U. The evolution of the conservative approach to breast cancer. Breast. 2007 Apr;16(2):120-9. doi: 10.1016/j.breast.2006.11.001. PMID 17403449
- [Background] Ciocca M, Pedroli G, Orecchia R, Guido A, Cattani F, Cambria R, Veronesi U. Radiation survey around a Liac mobile electron linear accelerator for intraoperative radiation therapy. J Appl Clin Med Phys. 2009 Apr 28;10(2):131-138. doi: 10.1120/jacmp.v10i2.2950. PMID 19458597
- [Background] Orecchia R, Ivaldi GB, Leonardi MC. Integrated breast conservation and intraoperative radiation therapy. Breast. 2009 Oct;18 Suppl 3:S98-102. doi: 10.1016/S0960-9776(09)70283-8. PMID 19914553
- [Background] Petit JY, Veronesi U, Orecchia R, Rey P, Martella S, Didier F, Viale G, Veronesi P, Luini A, Galimberti V, Bedolis R, Rietjens M, Garusi C, De Lorenzi F, Bosco R, Manconi A, Ivaldi GB, Youssef O. Nipple sparing mastectomy with nipple areola intraoperative radiotherapy: one thousand and one cases of a five years experience at the European institute of oncology of Milan (EIO). Breast Cancer Res Treat. 2009 Sep;117(2):333-8. doi: 10.1007/s10549-008-0304-y. Epub 2009 Jan 17. PMID 19152026
- [Background] Galimberti V, Ciocca M, Leonardi MC, Zanagnolo V, Paola B, Manuela S, Sahium RC, Lazzari R, Gentilini O, Peccatori F, Veronesi U, Orecchia R. Is electron beam intraoperative radiotherapy (ELIOT) safe in pregnant women with early breast cancer? In vivo dosimetry to assess fetal dose. Ann Surg Oncol. 2009 Jan;16(1):100-5. doi: 10.1245/s10434-008-0172-z. Epub 2008 Oct 21. PMID 18941842
- [Background] Rampinelli C, Bellomi M, Ivaldi GB, Intra M, Raimondi S, Meroni S, Orecchia R, Veronesi U. Assessment of pulmonary fibrosis after radiotherapy (RT) in breast conserving surgery: comparison between conventional external beam RT (EBRT) and intraoperative RT with electrons (ELIOT). Technol Cancer Res Treat. 2011 Aug;10(4):323-9. doi: 10.7785/tcrt.2012.500209. PMID 21728389
- [Result] Intra M, Luini A, Gatti G, Ciocca M, Gentilini OD, Viana AA, Chagas EM, Berrettini A, Schuh F, Scarpa D, Orecchia R, Veronesi U. Surgical technique of intraoperative radiation therapy with electrons (ELIOT) in breast cancer: a lesson learned by over 1000 procedures. Surgery. 2006 Sep;140(3):467-71. doi: 10.1016/j.surg.2006.03.019. No abstract available. PMID 16934611
- [Derived] Orecchia R, Veronesi U, Maisonneuve P, Galimberti VE, Lazzari R, Veronesi P, Jereczek-Fossa BA, Cattani F, Sangalli C, Luini A, Caldarella P, Venturino M, Sances D, Zurrida S, Viale G, Leonardi MC, Intra M. Intraoperative irradiation for early breast cancer (ELIOT): long-term recurrence and survival outcomes from a single-centre, randomised, phase 3 equivalence trial. Lancet Oncol. 2021 May;22(5):597-608. doi: 10.1016/S1470-2045(21)00080-2. Epub 2021 Apr 9. PMID 33845035
- [Derived] Veronesi U, Orecchia R, Maisonneuve P, Viale G, Rotmensz N, Sangalli C, Luini A, Veronesi P, Galimberti V, Zurrida S, Leonardi MC, Lazzari R, Cattani F, Gentilini O, Intra M, Caldarella P, Ballardini B. Intraoperative radiotherapy versus external radiotherapy for early breast cancer (ELIOT): a randomised controlled equivalence trial. Lancet Oncol. 2013 Dec;14(13):1269-77. doi: 10.1016/S1470-2045(13)70497-2. Epub 2013 Nov 11. PMID 24225155